CLINICAL TRIAL: NCT00996060
Title: A Phase 1 Protocol of Hydralazine and Valproic Acid in Advanced Solid Tumor Malignancies
Brief Title: Use of Hydralazine and Valproic Acid in Advanced Solid Tumor Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: New Mexico Cancer Research Alliance (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INST 0712C; NCI-2011-02651 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-03-26; First posted 2009-10-16 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2016-01

CONDITIONS: Lung Cancer
Keywords: Lung Cancer; Advanced Lung Cancer; Unresectable Lung cancer; Previously treated lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Hydralazine; Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hydralazine and Valproic Acid (Experimental): Starting dose of Hydralazine is 25 mg orally daily, days 1-28. (See Intervention for Dose Escalation Schema) Valproic acid 250 mg orally three times per day for days -14 through -8, then 500 mg orally three times per day daily for days -7 through 28, with the dose titrated to keep the serum level between 0.4 and 0.7 mM.
  Interventions: Drug: Hydralazine and Valproic Acid: Cohort -1; Drug: Hydralazine and Valproic Acid: Cohort 0; Drug: Hydralazine and Valproic Acid: Cohort 1; Drug: Hydralazine and Valproic Acid: Cohort 2; Drug: Hydralazine and Valproic Acid: Cohort 3; Drug: Hydralazine and Valproic Acid: Cohort 4; Drug: Hydralazine and Valproic Acid: Cohort 5

INTERVENTIONS:
Drug: Hydralazine and Valproic Acid: Cohort -1 — Initially, 3 patients will be enrolled into each cohort, beginning with the hydralazine 25 mg PO daily, with the valproic acid dosing beginning two weeks earlier to achieve a steady state level of valproic acid in the blood.
  In this cohort, Hydralazine is administered at 10 mg/day.
  Other Names: Depakote (Valproic Acid); Apresoline (Hydralazine)
Drug: Hydralazine and Valproic Acid: Cohort 0 — Initially, 3 patients will be enrolled into each cohort, beginning with the hydralazine 25 mg PO daily, with the valproic acid dosing beginning two weeks earlier to achieve a steady state level of valproic acid in the blood.
  Hydralazine is administered at 25 mg/day in this cohort.
  Other Names: Depakote (Valproic Acid); Apresoline (Hydralazine)
Drug: Hydralazine and Valproic Acid: Cohort 1 — Initially, 3 patients will be enrolled into each cohort, beginning with the hydralazine 25 mg PO daily, with the valproic acid dosing beginning two weeks earlier to achieve a steady state level of valproic acid in the blood.
  Hydralazine is administered at 50 mg/day in this cohort.
  Other Names: Depakote (Valproic Acid); Apresoline (Hydralazine)
Drug: Hydralazine and Valproic Acid: Cohort 2 — Initially, 3 patients will be enrolled into each cohort, beginning with the hydralazine 25 mg PO daily, with the valproic acid dosing beginning two weeks earlier to achieve a steady state level of valproic acid in the blood.
  Hydralazine is administered at 100 mg/day in this cohort as 25 mg four times per day.
  Other Names: Depakote (Valproic Acid); Apresoline (Hydralazine)
Drug: Hydralazine and Valproic Acid: Cohort 3 — Initially, 3 patients will be enrolled into each cohort, beginning with the hydralazine 25 mg PO daily, with the valproic acid dosing beginning two weeks earlier to achieve a steady state level of valproic acid in the blood.
  Hydralazine is administered at 200 mg/day in this cohort as 50 mg four times per day.
  Other Names: Depakote (Valproic Acid); Apresoline (Hydralazine)
Drug: Hydralazine and Valproic Acid: Cohort 4 — Initially, 3 patients will be enrolled into each cohort, beginning with the hydralazine 25 mg PO daily, with the valproic acid dosing beginning two weeks earlier to achieve a steady state level of valproic acid in the blood.
  Hydralazine is administered at 300 mg/day in this cohort as 75 mg four times per day.
  Other Names: Apresoline (Hydralazine); Depakote (Valproic Acid)
Drug: Hydralazine and Valproic Acid: Cohort 5 — Initially, 3 patients will be enrolled into each cohort, beginning with the hydralazine 25 mg PO daily, with the valproic acid dosing beginning two weeks earlier to achieve a steady state level of valproic acid in the blood.
  Hydralazine is administered at 400 mg/day in this cohort as 100 mg four times per day.
  Other Names: Apresoline (Hydralazine); Depakote (Valproic Acid)

SUMMARY:
1. Primary Objective:

   The primary endpoint to this study will be to document the toxicities, and reversibility of toxicities, of this regimen of hydralazine and valproic acid in patients with advanced, unresectable, previously treated lung cancers, for whom no acceptable standard therapy is available. A primary endpoint will be to determine any potential dose limiting toxicities, and the Maximal Tolerated Dose of this regimen.
2. Secondary Objectives:

The secondary endpoint of this study will be to determine any potential anti-tumor effects, as determined by the objective tumor response (complete and partial responses), clinical benefit (complete and partial responses, and clinical benefit), the time to tumor response, the time to tumor progression, and the overall survival.

DETAILED DESCRIPTION:
This study will be an open-label, non-randomized, dose-escalation phase I trial which will enroll in sequential cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. All patients with lung cancer who have disease which has been previously treated and/or for which there is no acceptable standard treatment regimen available, and cannot be treated definitively with either surgery or radiotherapy.
2. All will be appropriate candidates for treatment, and are not candidates for treatment with protocols of higher priority.
3. All patients should have an ECOG/Zubrod/SWOG performance status of less than 2 at the time of the initiation of therapy
4. Adequate end-organ function
5. No severe comorbid disease
6. Ability to provide informed consent.
7. Signed Informed Consent
8. ECOG/Zubrod/SWOG Performance Status less than 2
9. Life expectancy greater than 8 weeks
10. Male or female' age greater than 18 years
11. Patients of childbearing potential must be using an effective means of contraception.
12. Histologic diagnosis of lung cancer that is advanced and cannot be treated adequately by radiotherapy or surgery; or metastatic disease, and for which there is no standard chemotherapeutic option remaining or available
13. All participants must have either previously received or refused standard chemotherapy
14. Baseline laboratory values (bone marrow, renal, hepatic):

Adequate bone marrow function:

1. Absolute neutrophil count greater than 1000/µL
2. Platelet count greater than 100'000/µL

Renal function:

a. Serum creatinine less than 2.0 mg %

Hepatic function:

1. Bilirubin less than 1.5x normal
2. Serum calcium less than 12 mg/dl

Exclusion Criteria

1. Pregnant or lactating females
2. Myocardial infarction or ischemia within the 6 months before Cycle 0' Day 0
3. Uncontrolled' clinically significant dysrhythmia
4. Prior radiotherapy to an indicator lesion unless there is objective evidence of tumor growth in that lesion
5. Prior autoimmune disease
6. Uncontrolled metastatic disease of the central nervous system
7. Radiotherapy within the 2 weeks before Cycle 1' Day -14
8. Surgery within the 2 weeks before Cycle 1' Day -14
9. Any co morbid condition that' in the view of the attending physician' renders the patient at high risk from treatment complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2008-07; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
A primary endpoint will be to determine any potential dose limiting toxicities, & the Maximal Tolerated Dose of hydralazine & valproic acid regimen. | 28 days

SECONDARY OUTCOMES:
To determine any potential anti-tumor effects, as determined by the objective tumor response, clinical benefit, the time to tumor response, the time to tumor progression, and the overall survival. | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Monte Shaheen, M.D., Principal Investigator — University of New Mexico Cancer Center
Locations (1):
- University of New Mexico Cancer Center, Albuquerque, New Mexico, United States

REFERENCES:
- See also: University of New Mexico Cancer Center — http://www.cancer.unm.edu
- See also: New Mexico Cancer Care Alliance — http://www.nmcca.org